CLINICAL TRIAL: NCT06321536
Title: Response to Emerging Antimicrobial Resistance With Containment Microbiota Therapy
Brief Title: Response to Emerging Antimicrobial Resistance With Containment Microbiota Therapy (REACT)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Woodworth, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007230; U54CK000601 (NIH)
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Multi-Drug Resistant Organism Colonization
Keywords: Multi-Drug Resistant Organism; Fecal Microbiota Transplant; Antibiotic Resistance; Long-Term Care Facilities
MeSH Terms: interventions — Glycerol; Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: microbiota therapy (MT) (Experimental): Group 1 will offer Microbiome therapeutic (MT) to all MDRO-positive patients (i.e., intervention condition).
  Interventions: Drug: Allogeneic Microbiota in Glycerol (9%) (AMG)
- Group 2: Observation (No Intervention): Group 2 will be assigned to observation.

INTERVENTIONS:
Drug: Allogeneic Microbiota in Glycerol (9%) (AMG) — Participants will receive an Emory-manufactured MT product, delivered as 250mL via rectal enema or 30mL instillation via an existing functioning feeding tube with the rate adjusted to participant tolerance. Participants will receive three doses over the first seven days of the study.
  Other Names: Fecal Microbiota Transplant (FMT); Microbiome therapeutic (MT); Stool from healthy donors in saline suspension with 9% glycerol by volume
  Arms: Group 1: microbiota therapy (MT)

SUMMARY:
REACT is a phase two, open-label, randomized, controlled trial of microbiota therapy (MT) to reduce colonization with multi-drug resistant organisms (MDRO). REACT is designed to assess the safety and efficacy of MT administered to subjects colonized with a MDRO. The overarching hypothesis is that MT can reduce MDRO colonization with safety that is comparable to observation.

DETAILED DESCRIPTION:
REACT is a phase two, open-label, randomized, controlled trial of microbiota therapy (MT) to reduce colonization with multi-drug resistant organisms (MDRO) in patients admitted to long-term care facilities. REACT is designed to test the safety and efficacy of instillation of donor intestinal microbiota.

Patients admitted to long-term care facilities (e.g. long-term acute care hospitals and ventilator-capable skilled nursing facilities) found to be MDRO colonized during prevalence screening activities performed in the related APPS study.

Facilities undergo prevalence sampling that involves participant peri-rectal, inguinal, and stool sampling to estimate the prevalence of targeted MDROs (CRE, ESBL, VRE, MDRP) under the accompanying APPS protocol. Patients who are positive with at least one targeted MDRO are eligible for an Emory manufactured MT product (via rectal enema or feeding tube), or observation followed by repeat sampling at Days 7, 14, 21, and 28. Participants will be followed with collection of data on adverse events/safety/changes in medications at Days 0, 7, 14, 21, 28, and followed up once a month for 6 months, after MT administration.

ELIGIBILITY:
Inclusion Criteria:

1. Be able (or have available a Legal Authorized Representative who is able) to understand and sign a written informed consent document.
2. Be at least 18 years old at the time of consent.
3. Be able to comply with all study protocol requirements, including able to receive MT as retention enema or via enteral feeding tube and be available for the duration of the study follow up.
4. Be colonized with a target MDRO (CRE, VRE, ESBL, MDR Pseudomonas) as detected by bacterial culture of stool or peri-rectal swab (collected in companion APPS facility prevalence sampling protocol).
5. Be able to discontinue or complete planned courses of antibiotics, probiotics, and other microbiota restoration therapies by Day -1 and not resume until after Day 28.
6. The effects of the MT on the developing human fetus are unknown. For this reason, persons of child-bearing potential (POCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
7. Agree to refrain from receptive anal intercourse until the last biological specimen (stool sample or peri-rectal swab) is collected (Day 28).

Exclusion Criteria:

1. Are pregnant, breastfeeding, lactating, or planning a pregnancy during study duration (through 4 weeks after the last dose of investigational product, or MT), if POCBP.
2. Have known uncontrolled intercurrent illness(es):

   1. Symptomatic congestive heart failure
   2. Acute coronary syndrome
   3. Cardiac arrhythmia
   4. Untreated in-situ colorectal cancer
   5. Toxic megacolon
   6. Ileus
   7. Positive stool studies without completion of treatment course (including ova and parasites, Salmonella spp, Shigella, Campylobacter, and other enteropathogens).
   8. other acute illness that in the opinion of the investigator could affect the safety of the participant or make study data uninterpretable.
3. Are on systemic antibiotics for any reason other than treatment of recent MDRO infection or clear anticipated need for antibiotics during the follow up period that cannot be rescheduled (e.g. fluoroquinolone prophylaxis for percutaneous nephrostomy tube exchange, prolonged antibiotic course for endocarditis). Participants must complete the planned antibiotic course by study Day -1.
4. Have a compromised immune system, defined as:

   1. AIDS with CD4+ T-cell count <200 and detectable HIV viral load on most recent assay.
   2. Absolute neutrophil count (ANC) <1,000 neutrophils / mL on day of enrollment.
   3. Active malignancy requiring intensive induction chemotherapy, radiotherapy, or biologic treatment within 2 months prior to enrollment.
   4. History of hematopoietic cell transplantation, either allogeneic or autologous in the last 1 year.
5. Have a history of significant food allergy that led to anaphylaxis or hospitalization.
6. Have a life expectancy of 24 weeks or less
7. Have any condition that, in the opinion of the investigator, might interfere with study objectives or limit compliance with study requirements, including but not limited to:

   1. Known active intravenous drug or alcohol abuse
   2. Uncontrolled psychiatric illness
   3. Social situations (e.g. incarceration)
8. Received an interventional agent (drug, device, or procedure) within 28 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference in number of solicited Adverse Events (AEs) | Day 0, Day 7 post-intervention
  Difference in number of solicited AEs between Day 0 and Day 7 in AMG-treated vs Observation participants.
Difference in severity of solicited AEs | Day 0, Day 7 post-intervention
  Difference in severity of solicited AEs will be compared in AMG-treated vs Observation participants. Graded as mild, moderate or severe, up to 7 days post-intervention.
Difference in number of unsolicited AEs | Day 0, Day 28 post-intervention
  Difference in number of unsolicited AEs between Day 0 and Day 28 in AMG-treated vs Observation participants.
Difference in severity of unsolicited AEs | Day 0 and Day 28
  Difference in severity of unsolicited AEs will be collected between Day 0 and Day 28. Graded as mild, moderate or severe and compared in AMG-treated vs Observation participants
Difference in proportion of participant stool positive cultures for any target MDRO among AMG-treated compared to Observation participants | Day 28 post-intervention
  Difference in proportion of participant stool cultures at Day 28 positive will be measured for any target MDRO among AMG-treated compared to Observation participants

SECONDARY OUTCOMES:
Count of serious AEs (SAEs) | Day 180
  Count of serious AEs (SAEs) between Day 0 and Month 6 (Day 180) censored by last telephone visits or death, whichever is later.
Count of AEs of Special Interest (AESIs) | Day 180
  Count of AEs of Special Interest (AESIs) at day Day 180, censored by last telephone visit or death, whichever is later.
Proportion of stool cultures at Day 28 positive for category-specific MDROs | Day 28
  Proportion of stool cultures at Day 28 positive for category-specific MDROs (e.g. ESBL, CRE, MDRP, VRE).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Woodworth, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - A.G Rhodes Wesley Woods, Atlanta, Georgia
  - Emory Long Term Acute Care (LTAC), Decatur, Georgia
  - RML Specialty Hospital, Hinsdale, Illinois
  - Penn Medicine Rittenhouse, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant solicited adverse event and serious adverse event data will be shared.
  Isolate genomic data and participant metagenomic data will be shared in public repositories (NCBI) at time of publication
Supporting Information: Study Protocol
Time Frame: Data will become available at time of publication.
Access Criteria: Sequence data access will not be restricted. Additional participant-level data will be shared by review of PI of proposing investigators and appropriate ethical approval (e.g. IRB) if any.